CLINICAL TRIAL: NCT07285148
Title: An Open-label, Multicenter Phase Ib/II Study to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of ANS014004 in Combination With EGFR-TKI in Patients With EGFR Mutation-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate ANS014004 in Combination With EGFR-TKI in Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Collaborators: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANS014004/PLB1004NSCLC-IbII-01
Record Dates: First submitted 2025-11-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; EGFR Mutation; Metastatic Lung Cancer; MET Alteration
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANS014004+PLB1004 (Experimental): The Phase Ib study consists of two parts: dose escalation and dose optimization. The dose escalation part will enroll participants with EGFR mutation-positive locally advanced or metastatic NSCLC who have received prior standard therapy in order to evaluate the safety and tolerability of the combination therapy and determine the maximum tolerated dose (MTD) (if any); The dose optimization part will further expand the population to include participants with EGFR mutation-positive locally advanced or metastatic NSCLC who have not received prior systemic therapy for advanced disease or have received standard therapy to determine the recommended Phase 2 dose (RP2D).
  Interventions: Drug: ANS014004 + PLB1004
- ANS014004 + Osimertinib (Active Comparator): participants will be enrolled in into two cohorts according to the prior anti-tumor treatment received.
  * Cohort A: participants with EGFR mutation-positive (excluding exon 20 insertions) locally advanced or metastatic NSCLC who have not received prior standard systemic therapy for advanced disease. Participants who meet the inclusion criteria will be stratified according to baseline brain metastasis status (present vs. absent) and be randomized at a ratio of 2:1 to receive the combination treatment of ANS014004 and PLB1004 or the combination treatment of ANS014004 and Osimertinib.
  * Cohort B: participants with EGFR mutation-positive (excluding exon 20 insertions) locally advanced or metastatic NSCLC who previously received standard systemic therapy. Participants who meet the inclusion criteria will be stratified according to baseline MET amplification and/or overexpression status (present vs. absent) and be randomized at a ratio of 2:1 to receive the combination treatment of ANS0140
  Interventions: Drug: ANS014004 + Osimertinib

INTERVENTIONS:
Drug: ANS014004 + PLB1004 — 1. Drug: ANS014004 Investigational Type II MET tyrosine kinase inhibitor (oral tablets). Dosing: Phase Ib escalation (30 mg, 45 mg, 60 mg, 75 mg QD); optimization uses selected doses; Phase II uses RP2D. Administered QD (≥1h before/2h after meals) in 21-day cycles. Targets MET exon 14 skipping, amplification, overexpression, and fusions.
  2. Drug: PLB1004 Investigational irreversible EGFR tyrosine kinase inhibitor (oral capsules). Fixed dose: 80 mg QD. Administered QD (≥1h before/2h after meals) in 21-day cycles. Targets EGFR classical mutations (Ex19del, L858R), rare mutations, Ex20ins, and T790M.
  Arms: ANS014004+PLB1004
Drug: ANS014004 + Osimertinib — 1. Drug: ANS014004 (Same description as above, as the drug is identical across arms).
  2. Drug: Osimertinib Market-approved third-generation EGFR tyrosine kinase inhibitor (oral tablets). Dosing: Per reference label (QD, with/without meals). Administered in 21-day cycles. Targets EGFR classical mutations (Ex19del, L858R) and T790M. Used as an active comparator.
  Arms: ANS014004 + Osimertinib

SUMMARY:
Protocol Title

A Study to Evaluate ANS014004 in Combination with EGFR-TKI in Patients with EGFR Mutation-Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer

The main purpose of this research study is to

Find a safe and tolerable dose of two investigational drugs, ANS014004 and PLB1004, when used together.

Learn how effective this drug combination is at treating a type of lung cancer called "EGFR mutation-positive non-small cell lung cancer (NSCLC)" that has spread to other parts of the body (locally advanced or metastatic).

This study is trying to answer the following questions:

Safety & Dosing: What are the side effects of combining ANS014004 and PLB1004? What is the best dose to use that patients can tolerate well?

Effectiveness: Can this combination of drugs help shrink patients' tumors or stop them from growing?

Background Information

For patients with advanced lung cancer that has a specific gene change called an "EGFR mutation," targeted therapies known as EGFR-TKIs are a standard treatment. While these treatments often work well at first, most tumors eventually stop responding to the drug (this is called "acquired resistance"). The investigational drug ANS014004 is designed to block a protein called MET, which is one of the ways that tumors become resistant to EGFR-TKIs. The researchers believe that by combining ANS014004 with the EGFR-TKI PLB1004, they may be able to prevent or delay resistance, offering patients a more effective and longer-lasting treatment option.

How will the study be conducted?

This study is divided into two parts:

Part 1 (Dose Escalation and Optimization): A small number of participants will receive different dose levels of ANS014004 combined with a fixed dose of PLB1004. The goal is to find the safest and most tolerable dose combination.

Part 2 (Phase II Study): Once a recommended dose is identified, more participants will be enrolled to further evaluate how well the drug combination works against the cancer.

Throughout the study, participants' health will be closely monitored, and their tumors will be measured regularly using imaging scans (like CT scans) to see how they respond to the treatment.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Male or female participants ≥18years of age at the time of signing the informed consent form.
2. Patients with histologically or cytologically confirmed diagnosis of unresectable locally advanced (Stage IIIB and IIIC) or metastatic (Stage IV) NSCLC (according to the lung cancer staging criteria, refer to the eighth edition of the American Joint Committee on Cancer [AJCC] Lung Cancer Staging).
3. Have a documented EGFR positive mutation (EGFR classic mutations including ex19del and ex21 L858R, uncommon mutations and ex20 insertion mutations) in tumor tissue samples or pleural fluid or blood samples.
4. For Phase Ib dose escalation: have disease progression after the existing standard of care or intolerance to the existing standard of care or inappropriate or no effective standard of care is available (standard of care is defined as treatment recommended by the National Comprehensive Cancer Network [NCCN] guidelines [including but not limited to chemotherapy, radiotherapy, targeted therapy based on mutation status, immunotherapy, and surgery]). For participants who are considered intolerant to or ineligible for available standard therapy, or for whom effective standard therapy does not exist, the documentation of these reasons is required.

   For Phase Ib dose optimization and Phase II study: have or haven't received prior standard systemic therapy for advanced disease.

   Standard systemic therapy is referred to as (country-specific approved treatment will also be applied):
   * EGFR classic mutations: EGFR-TKIs alone or in combination (examples, gefitinib and osimertinib with or without chemotherapy) for ex19del and ex21 L858R. Osimertinib or other third-generation EGFR TKI for T790M mutation.
   * EGFR uncommon mutations: EGFR-TKIs or chemotherapy for uncommon mutations including but not limited to G719X, S768I, L861Q mutations.
   * EGFR exon 20 activating insertions: chemotherapy with or without amivantamab or country-specific approved EGFR TKIs.
5. For China only: the presence of MET amplification and/or overexpression in tumor tissue samples or pleural fluid or blood samples collected after progression on prior EGFR-TKI treatment, confirmed by a central /local laboratory.

   MET amplification is defined as the presence of MET amplification confirmed by nextgeneration sequencing (NGS) technology or mean MET gene copy number (GCN) ≥ 4 per cell or the ratio of MET to chromosome enumerating probe against chromosome 7 (MET/CEP7) ≥2.0 confirmed by fluorescence in situ hybridization (FISH) testing.

   MET overexpression is defined as immunohistochemistry (IHC) ≥ 2+ (local or central lab test results are accepted).
6. Have at least one measurable target lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
7. ECOG PS ≤ 1.
8. Life expectancy of ≥12 weeks, in the opinion of the investigator.
9. Adequate organ function as determined by medical evaluation (within 7 days prior to study treatment) including:

   * Adequate hematologic status, defined as: absolute neutrophil count (ANC) ≥1.5×109/L, hemoglobin ≥90 g/L, platelets ≥75×109/L. Platelet transfusions are not permitted within 3 days, red blood cell transfusions are not permitted within 14 days, hematopoietic growth factors are not permitted within 7 days (14 days for PEGylated granulocyte colony stimulating factor [G-CSF] or erythropoietin) prior to obtaining these laboratory values.
   * Adequate hepatic function, defined as: serum TBIL ≤1.5× ULN (in participants with known Gilbert's syndrome, TBIL ≤3× ULN with direct bilirubin ≤1.5× ULN), serum ALT or AST ≤2.5× ULN (or 5.0× ULN for documented liver metastasis).
   * Adequate renal function, defined as: creatinine clearance ≥60 mL/min (calculated by Cockcroft-Gault formula or CKD EPI formula [Appendix 4 of Section 12.4]).
   * Adequate coagulation profile, defined as (including if receiving anticoagulant therapy):

   prothrombin time (PT)< 1.5 × ULN, activated partial thromboplastin time (APTT)< 1.5 × ULN. If the participant is on anticoagulant therapy, must be on a stable dose of anticoagulant for at least1month prior to the study treatment.
10. Female participants should be using adequate contraceptive measures until 90 days after the EOT, should not be breast feeding and must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test within 7 days prior to start of dosing if of childbearing potential; or must have evidence of non-child bearing potential by fulfilling one of the following criteria at screening.

    * Achieved postmenopausal status, refer to NCCN Guidelines for Breast Cancer (2024V3.0) for the detailed definition of menopause.
    * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
11. Male participants of childbearing potential are required to use adequate contraception (i.e., barrier method of birth control), during their participation in the study and for 90 days following the EOT. Male participants must also refrain from donating sperm during their participation in the study and for 90 days following the last dose of study treatment.
12. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this study.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Have other known primary driver gene alterations. For example, NSCLC with a targetable alteration in ALK, RET, ROS1, BRAF, KRAS, etc. The investigators should discuss enrollment with the sponsor regarding co-mutations.
2. Prior treated with hepatocyte growth factor (HGF) targeted therapy or other MET-TKIs (including Type I and Type II), e.g., gulmonertinib, savolitinib, capmatinib, tepotinib, bozitinib, cabozantinib, glenitinib and almonertinib.
3. Participation in other therapeutic clinical trials within 28 days prior to the first dose of study treatment.
4. Received anti-tumor therapy (chemotherapy, immunotherapy, hormone therapy, targeted therapy, biological therapy or other anti-tumor therapy, except for hormones for hypothyroidism or estrogen replacement therapy, anti-estrogen analogs, and agonists required to inhibit serum testosterone levels) within 14 days or 5 half-lives (whichever is shorter) of the first dose of study treatment. The following exceptions are:

   * Nitrosourea or mitomycin-C within 6 weeks prior to the first dose of study treatment.
   * Chinese medicines with anti-tumor indications within 7 days prior to the first dose of study treatment.
5. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days of the first dose of study treatment.

   Participants must have recovered from all radiation related toxicity, not requiring corticosteroids.
6. Major surgery, other than diagnostic surgery, within 4 weeks of the first study treatment or is expected during the study.
7. Toxicities of prior therapy have not been resolved to Grade ≤1 or to baseline, as evaluated by NCI-CTCAE v5.0. NOTE: Participants with Grade 2 toxicities can be enrolled if the toxicities as stable and do not affect the safety of participating in this study (e.g., alopecia, skin hyperpigmentation, neuropathy).
8. History of another primary malignancy that has been diagnosed or required therapy within the past 3 years (other than adequately treated local basal cell or squamous cell carcinoma of the skin; or any other cancer in situ currently in complete remission).
9. Have central nervous system (CNS) metastases that are symptomatic or clinically unstable or require increased steroid dose to manage CNS symptoms within 4 weeks prior to the first dose of study treatment.

   * Participants with symptomatic CNS metastases may participate in the study providing that symptoms are controlled after treatment, clinically stable for at least 4 weeks and have no evidence of new or enlarged brain metastases.
   * Participants with carcinomatous meningitis or meningeal metastases, or spinal cord compression are excluded regardless of clinical stability.
   * Participants with asymptomatic CNS metastases with a maximum diameter of brain metastases <3 cm by imaging (such as MRI) without significant cerebral edema are eligible for the study.
10. Participants with clinically uncontrollable third-space effusion, including but not limited to pleural effusion, peritoneal effusion or pericardial effusion, are assessed by the investigator to be unsuitable for the study treatment.
11. Participants receiving unstable or increasing doses of corticosteroids. For participants receiving corticosteroids for endocrine deficiencies or symptoms associated to their disease (excluding CNS disease), the dose must have been stabilized (or reduced) for at least 14 days before the first dose of study treatment.
12. Have a history of or ongoing severe retinopathy.
13. Presence of serious cardiovascular or cerebrovascular disease, including but not limited to:

    * Mean resting corrected QT interval corrected by Fridericia's formula (QTcF) >470 msec obtained from triplicate 12-lead electrocardiograms (ECGs).
    * Symptomatic heart failure per New York Heart Association (NYHA) classification Class II or above.
    * Baseline left ventricular ejection fraction (LVEF) below institution's lower limit of normal (LLN) or <50% if assessed by echocardiography (ECHO) or Multigated Radionuclide Angiography (MUGA).
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, third degree heart block, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
    * Presence of any factors that increase the risk of QTc prolongation or the risk of arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or use of any concomitant medication known to prolong the QT interval within 14 days prior to the first dose of study treatment.
    * Any of the following within 6 months prior to the first dose of the study treatment: myocardial infarction, severe/unstable angina, coronary artery bypass graft, congestive heart failure, cardiomyopathy, pulmonary embolism, cerebrovascular accident, or transient ischemic attack.
14. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including but not limited to:

    * Uncontrolled hypertension, defined as a systolic blood pressure (BP) ≥160 mmHg or diastolic BP ≥100 mmHg despite medical therapy. Participant with a history of hypertension is allowed if BP is stable and controlled within these limits by antihypertensive treatment.
    * Previous history of, or presence of clinically symptomatic or at high risk for interstitial lung disease or interstitial pneumonitis, including radiation pneumonitis (i.e., affecting activities of daily living or requiring therapeutic treatment).
    * Unstable or uncompensated respiratory and renal disease, active bleeding diseases.
15. Uncontrolled concurrent infection including but not limited to:

    * Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

      * If hepatitis B surface antigen (HBsAg) is positive, HBV DNA assay should be performed. Participants may be eligible if HBV DNA test value ≤ ULN.
      * If HCV antibody is positive, HCV ribonucleic acid (RNA) assay should be performed. Participants may be eligible if HCV RNA negative.
    * Known human immunodeficiency virus (HIV) infection or known history of acquired immunodeficiency syndrome (AIDS).
    * Syphilis positive.
    * Active tuberculosis infection.
    * Onset period of keratitis or ulcerative keratitis.
    * Other active infections requiring systemic treatment within 14 days prior to the first dose of study treatment.
16. Unwilling or unable to comply with the requirements of oral drug administration, or presence of gastrointestinal disorders such as refractory nausea and vomiting, any acute or chronic gastrointestinal disorder, inability to swallow the formulation, or prior major bowel resection that may prevent adequate absorption of ANS014004 or PLB1004.
17. Hypersensitivity to ANS014004, PLB1004 or their excipients, or history of allergic reactions to ANS014004 and PLB1004 with similar chemical or biological structure or similar drugs.
18. Concomitant use of drugs metabolized by P-glycoprotein (P-gp)/breast cancer resistance protein (BCRP) or OCT2/OATP1B1/MATE1, or moderate or strong inducers or inhibitors of P-gp/BCRP or CYP2B6/CYP2C9/CYP2C19/OCT2/OATP1B1/MATE1 within 5 half-lives before the use of the study treatment. For dose escalation part only: concomitant treatment with moderate or strong P-gp/BCRP or CYP2C8/CYP2D6/CYP3A4 inducers or inhibitors within 5 half-lives prior to administration of study treatment.
19. In receipt of any live attenuated vaccination within 30 days prior to the first dose of study therapy.
20. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
21. Have prior or ongoing clinically significant illness, medical condition, surgical history, physical findings, or laboratory abnormality that, in the investigator's opinion, would not be in the best interest of the participant; or that could alter the absorption, distribution, metabolism, or excretion of the study treatment; or impair the assessment of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity (DLT) during the DLT observation period (Phase Ib Dose Escalation) | 2 years.
  To evaluate the tolerability of ANS014004 in combination with PLB1004. DLT is defined per NCI-CTCAE v5.0 (e.g., Grade 4 neutropenia lasting ≥7 days, febrile neutropenia, Grade 4 thrombocytopenia, Hy's Law-meeting hepatotoxicity, Grade ≥3 non-hematologic/non-hepatic toxicity excluding specified exceptions, etc.). The DLT observation period is the first 28 days after treatment initiation (including single-dose period and Cycle 1 of multiple-dose period). The outcome will be reported as the count and proportion of participants experiencing DLT in each dose group.
Maximum tolerated dose (MTD) of ANS014004 in combination with PLB1004 (Phase Ib Dose Escalation) | 2 years
  To determine the MTD of the combination therapy. MTD is defined as the highest dose level where ≤1 of 3-6 evaluable participants experience DLT during the DLT observation period. The outcome will be reported as the specific dose of ANS014004 (e.g., 45 mg QD, 60 mg QD) combined with fixed 80 mg QD PLB1004 that meets the MTD definition.
Objective Response Rate (ORR) assessed by investigator per RECIST v1.1 (Phase Ib Dose Optimization, Phase II) | 2 years
  To evaluate the anti-tumor activity of ANS014004 in combination with PLB1004 (Phase Ib Dose Optimization) or ANS014004 combined with PLB1004/Osimertinib (Phase II) in EGFR mutation-positive locally advanced or metastatic NSCLC. ORR is defined as the proportion of participants with confirmed Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Tumor assessments are performed every 6 weeks (±7 days) for the first year and every 12 weeks (±7 days) thereafter. The outcome will be reported as the proportion of participants achieving ORR, with 95% confidence intervals (CIs) calculated using the Clopper-Pearson method.
Recommended Phase 2 Dose (RP2D) of ANS014004 in combination with PLB1004 (Phase Ib Dose Optimization) | 2 years.
  To identify the RP2D of the combination therapy. RP2D is determined based on comprehensive analysis of safety (incidence of AEs/DLTs), pharmacokinetic (PK) data, and preliminary efficacy (ORR, DCR) from the Phase Ib Dose Optimization period. The outcome will be reported as the specific dose of ANS014004 (e.g., 60 mg QD) combined with fixed 80 mg QD PLB1004 selected for Phase II.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) assessed by NCI-CTCAE v5.0 (All Phases) | 2 years
  To evaluate the safety/tolerability of ANS014004 combinations. AEs include treatment-related AEs (TRAEs), serious AEs (SAEs), and AEs leading to dose modification/discontinuation. Severity is graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0 (Grade 1-5). AEs are collected from the first dose of study treatment to 28 days after the last dose or before new anti-tumor treatment. The outcome will be reported as the count and proportion of participants with AEs by severity, system organ class (SOC), and preferred term (PT).
Plasma maximum observed concentration (Cmax) of ANS014004 (All Phases) | 2 years
  To characterize the PK profile of ANS014004 in combination with PLB1004/Osimertinib. Cmax is defined as the highest plasma concentration of ANS014004 measured after drug administration. PK blood samples are collected at pre-specified time points (e.g., pre-dose, 0.5h, 1h, 2h, 4h, 6h, 8h, 10h, 24h post-dose in Phase Ib Dose Escalation). The outcome will be reported as descriptive statistics (arithmetic mean, geometric mean, standard deviation, minimum, maximum) of Cmax by study phase and dose group.
Plasma area under the concentration-time curve from time 0 to last quantifiable time point (AUC0-t) of ANS014004 (All Phases) | 2 years
  To characterize the PK profile of ANS014004. AUC0-t is defined as the area under the plasma concentration-time curve of ANS014004 from time 0 to the last time point with a quantifiable concentration. PK samples are collected per pre-specified schedules (e.g., Table 3-5 in the protocol). The outcome will be reported as descriptive statistics (arithmetic mean, geometric mean, coefficient of variation) of AUC0-t by study phase and dose group.
Disease Control Rate (DCR) assessed by investigator per RECIST v1.1 (Phase Ib Dose Optimization, Phase II) | 2 years
  To evaluate the anti-tumor efficacy of ANS014004 combinations. DCR is defined as the proportion of participants with confirmed CR, PR, or Stable Disease (SD) per RECIST v1.1. Tumor assessments follow the same schedule as ORR (every 6 weeks for the first year, every 12 weeks thereafter). The outcome will be reported as the proportion of participants achieving DCR, with 95% CIs.
Duration of Response (DoR) assessed by investigator per RECIST v1.1 (Phase Ib Dose Optimization, Phase II) | 2 years
  To evaluate the durability of anti-tumor response. DoR is defined as the time from the first documentation of CR/PR to the first documentation of disease progression (PD) or death from any cause. The outcome will be reported as median DoR with 95% CIs, calculated using the Kaplan-Meier method.
Progression-Free Survival (PFS) assessed by investigator per RECIST v1.1 (Phase Ib Dose Optimization, Phase II) | 2 years
  To evaluate the time to disease progression or death. PFS is defined as the time from the first dose of study treatment to the first documentation of PD (per RECIST v1.1) or death from any cause. The outcome will be reported as median PFS with 95% CIs, using the Kaplan-Meier method.
Overall Survival (OS) (Phase Ib Dose Optimization, Phase II) | 2 years
  To evaluate the overall survival of participants. OS is defined as the time from the first dose of study treatment to death from any cause. Participants alive at the last follow-up are censored at the date of last known survival. The outcome will be reported as median OS with 95% CIs, using the Kaplan-Meier method.
Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) score (All Phases) | 2 years
  To evaluate overall disease-related symptoms via participant-reported outcomes (PROs). The NSCLC-SAQ is a validated questionnaire specific to NSCLC symptoms (e.g., cough, dyspnea, fatigue). Scores are collected at screening, Cycle 1 Day 1, Cycle 2 Day 1, every 6 weeks thereafter, end-of-treatment (EOT), and 28 days after last dose. The outcome will be reported as mean (±standard deviation) changes in NSCLC-SAQ scores from baseline to each time point.
Functional Assessment of Chronic Illness Therapy (FACIT) GP5 question score (All Phases) | 2 years
  To evaluate overall side effect impact and physical function via PROs. The GP5 question from the FACIT item library assesses the impact of treatment side effects on daily function (scored on a 0-4 scale, with higher scores indicating greater impact). Scores are collected at the same time points as NSCLC-SAQ. The outcome will be reported as mean (±standard deviation) changes in GP5 scores from baseline to each time point.
Plasma time to maximum observed concentration (Tmax) of ANS014004 (All Phases) | 2 years
  To characterize the PK profile of ANS014004. Tmax is defined as the time from drug administration to the first occurrence of Cmax. PK samples are collected per pre-specified schedules. The outcome will be reported as median (range) of Tmax by study phase and dose group.
Plasma half-life (t1/2) of ANS014004 (All Phases) | 2 years
  To characterize the PK profile of ANS014004. t1/2 is defined as the time required for the plasma concentration of ANS014004 to decrease by half. It is calculated via non-compartmental analysis (NCA) using Phoenix WinNonlin software. The outcome will be reported as mean (±standard deviation) of t1/2 by study phase and dose group.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center David H, Koch Center lor Cancer Care, New York, New York, United States